CLINICAL TRIAL: NCT00207688
Title: A Multicenter International Study of the Long-term Safety of Infliximab (REMICADE) in Ulcerative Colitis
Brief Title: A Long Term Safety Study of Infliximab (Remicade) in in Ulcerative Colitis Patients
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Janssen Biologics BV (Unknown)
Responsible Party: Sponsor
Other Study IDs: CR004801; C0168T62 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Infliximab; Remicade; Safety
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (3):
- Infliximab 5 mg/kg: This is an observational study which includes patients from primary studies C0168T37, C0168T46, C0168T72.
  Interventions: Drug: Infliximab 5 mg/kg
- Infliximab 10 mg/kg: This is an observational study which includes patients from primary studies C0168T37, C0168T46, C0168T72.
  Interventions: Drug: Infliximab 10 mg/kg
- Placebo: This is an observational study which includes patients from primary studies C0168T37, C0168T46, C0168T72.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Infliximab 5 mg/kg — Patients who received infliximab 5 mg/kg from C0168T37, C0168T46, C0168T72 studies will be observed.
  Groups: Infliximab 5 mg/kg
Drug: Infliximab 10 mg/kg — Patients who received infliximab10 mg/kg from C0168T37, C0168T46, C0168T72 studies will be observed.
  Groups: Infliximab 10 mg/kg
Drug: Placebo — Patients who received placebo from C0168T37, C0168T46, C0168T72 studies will be observed.
  Groups: Placebo

SUMMARY:
The purpose of this study is to evaluate long-term safety information of infliximab in patients who have participated in infliximab clinical studies in ulcerative colitis.

DETAILED DESCRIPTION:
This is a long term, multicenter, international safety study to evaluate targeted long-term safety information on patients who have participated in infliximab(Remicade) clinical studies in ulcerative colitis that require long-term safety follow-up. All patients who received at least one dose of study drug (infliximab or placebo) in the primary studies (C0168T37 ,C0168T46, C0168T72) are eligible to participate in this long-term safety follow-up study (C0168T62). Patients will begin participation in C0168T62 at the time of their last safety visit in the primary study and will be followed for 5 years. No study agent will be administered. Information on deaths, serious infections, new malignancies (including colorectal cancer) and new autoimmune diseases and surgical procedures (including colectomy) and hospitalizations for the treatment of ulcerative colitis will be collected. Information about possible delayed allergic reactions (possible fever, rash, fatigue, joint pain) will also be collected if patients received infliximab after the end of the primary study. In addition, data on dysplasia of the colon will be collected from patients who were identified in the primary study to be at high-risk for colon cancer and were required per protocol to undergo a follow-up colonoscopy as part of long-term safety follow-up. All adverse events, including non-serious adverse events, will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled in three Phase 3 Janssen-sponsored (C0168T37, C0168T46, C0168T72) infliximab clinical studies in ulcerative colitis that require long-term safety follow-up
* Patients must have received at least 1 dose of study agent to be eligible for participation in the study

Exclusion Criteria:

- Patients who refuse consent or are unwilling to respond to requests for long-term safety information within the required timeframe will be excluded. In addition, patients participating in a study extension to the primary study are not eligible for participation in the C0168T62 study during the study extension participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ulcerative colitis who have participated in infliximab clinical studies and must have received at least 1 dose of study medication to be eligible for participation in C0168T62.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2004-08-31 (Actual); Primary Completion 2015-09-09 (Actual); Study Completion 2015-09-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety | 5 years
  Long-term safety will be evaluated by assessment of serious infections,new malignancies (including colorectal cancer), new autoimmune diseases, death, delayed hypersensitivity (serum sickness-like) reactions, or dysplasia of the colon and other non-serious adverse events. Non-serious adverse events will be collected for participants continuing at the beginning of collection of non-serious adverse events.

SECONDARY OUTCOMES:
Number of patients with malignancies by malignancy type | 5 years
  Number of patients with malignancies by malignancy type (ie, lymphoma, nonmelanoma skin cancers, other malignancies)
Number of patients with serious infections by type of infection | 5 years
Number of patients with surgical procedures (including colectomy) for the treatment of ulcerative colitis | 5 years
Number of patients with hospitalizations for the treatment of ulcerative colitis | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (102):
- United States (44):
  - Scottsdale, Arizona
  - Anaheim, California
  - Los Angeles, California
  - Oakland, California
  - Orange, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Orlando, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Metairie, Louisiana
  - Laurel, Maryland
  - Boston, Massachusetts
  - Plymouth, Minnesota
  - Rochester, Minnesota
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Egg Harbor, New Jersey
  - Great Neck, New York
  - New Hyde Park, New York
  - New York, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Beaver Falls, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Memphis, Tennessee
  - Houston, Texas
  - Burlington, Vermont
  - Charlottesville, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Federal, Argentina
- Australia (8):
  - Bedford
  - Box Hill
  - Garran
  - Herston
  - Kogarah
  - Parkville
  - Perth
  - South Brisbane
- Austria (2):
  - Innsbruck
  - Vienna
- Belgium (4):
  - Antwerp
  - Brussels
  - Imeldalaan 9
  - Leuven
- Canada (10):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Edmonton
  - Halifax
- Czechia (2):
  - Pardubice
  - Prague
- Denmark (4):
  - Aalborg
  - Aarhus C
  - Copenhagen
  - Hvidovre
- France (5):
  - Lille
  - Nancy
  - Paris
  - Strasbourg
  - Toulouse
- Germany (3):
  - Berlin
  - München
  - Stade
- Israel (4):
  - Jerusalem
  - Kfar Saba
  - Rehovot
  - Tel Aviv
- Netherlands (3):
  - Eindhoven
  - Nijmegen
  - Rotterdam
- New Zealand (2):
  - Auckland
  - Christchurch
- Switzerland (3):
  - Basel
  - Bern
  - Zurich
- United Kingdom (7):
  - Cardiff
  - Dundee
  - Glasgow
  - Harrow
  - Liverpool
  - London
  - Manchester

REFERENCES:
- [Derived] Sandborn WJ, Rutgeerts P, Feagan BG, Reinisch W, Olson A, Johanns J, Lu J, Horgan K, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Colectomy rate comparison after treatment of ulcerative colitis with placebo or infliximab. Gastroenterology. 2009 Oct;137(4):1250-60; quiz 1520. doi: 10.1053/j.gastro.2009.06.061. Epub 2009 Jul 28. PMID 19596014
- See also: Multicenter International Study of the Long-term Safety of Infliximab (REMICADE®) in Ulcerative Colitis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=157&filename=CR004801_CSR.pdf